CLINICAL TRIAL: NCT03871088
Title: N-3 Fatty Acids as the First-line Antidepressant Therapy: From Biomarkers to Clinical Subtypes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Science and Technology Council, Taiwan (Other Government)
Responsible Party: Principal Investigator, Kuan-Pin, Professor, National Science and Technology Council, Taiwan
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: NHRI-EX105-10528NI
Record Dates: First submitted 2019-03-07; First posted 2019-03-12 (Actual); Last update posted 2019-03-12 (Actual); Status verified 2019-03

CONDITIONS: Major Depressive Disorder
Keywords: Depression, omega-3 fatty acids, nutritional intervention
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — Fatty Acids, Omega-3

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Eicosapentaenoic acid (EPA) (Active Comparator): Eicosapentaenoic acid (EPA) is an omega-3 fatty acid. In physiological literature, it is given the name 20:5(n-3).
  Interventions: Dietary Supplement: Omega-3 fatty acids
- Docosahexaenoic acid (DHA) (Experimental): Docosahexaenoic acid (DHA) is an omega-3 fatty acid. In physiological literature, it is given the name 22:6(n-3).
  Interventions: Dietary Supplement: Omega-3 fatty acids
- EPA/DHA combination (Active Comparator): EPA/DHA means the combination of omega-3 fatty acids Eicosapentaenoic and Docosahexaenoic acids.
  Interventions: Dietary Supplement: Omega-3 fatty acids

INTERVENTIONS:
Dietary Supplement: Omega-3 fatty acids — 12-week double-blind, randomized controlled trial

SUMMARY:
Investigate the clinical subtypes and the biological markers to personalize the use n-3 PUFAs (EPA, DHA, and EPA/DHA) in MDD.

DETAILED DESCRIPTION:
In this proposal, the investigators aim to explore the clinical subtypes and biological markers to personalize the use n-3 PUFAs (EPA, DHA, and EPA/DHA) in MDD. By stratifying the subjects with (versus without) remission and treatment response, the biological markers are expected to have important prediction effects in future clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* the diagnostic criteria of DSM-IV for MDD
* 18 to 65 years old
* pre-study ratings of 18 or greater on the 21-item Hamilton Rating Scale for Depression (HAMD)
* physically healthy under comprehensive evaluations in medical history, physical examination, and laboratory parameters tests
* have not received any psychiatric treatment in 2 weeks
* competent to receive a full explanation of this study and give written informed consent.

Exclusion Criteria:

* a recent or past history of other DSM-IV AxisI diagnoses besides unipolar major depression, including psychotic disorders, organic mental disorders, impulse control disorders, substance use disorder or substance abuse (last 6 months prior to the study), and bipolar disorders
* AxisII diagnoses, including borderline and antisocial personality disorder
* a notable medical comorbidity
* acutely suicidal ideation and attempt were noted that close monitoring such as hospitalization is necessary
* regular consumption of omega-3 PUFAs supplements or a habit of eating ﬁsh equal or more than 4 times per week

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2018-06 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Hamilton Rating Scale for Depression (HAMD) Changes | From Week 0 to Week 12
  The Changes of scores in Hamilton Rating Scale for Depression

SECONDARY OUTCOMES:
Response rate | at Week 12
  50% decreases in the Hamilton Rating Scale for Depression from W0 to W12
Remission rate | at Week 12
  Less than 8 points in the Hamilton Rating Scale for Depression at W12

CONTACTS AND LOCATIONS:
Locations (1):
- China Medical University Hospital, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: No